CLINICAL TRIAL: NCT07073898
Title: Population Health Management Approaches to Increase Lung Cancer Screening in Community Health Centers - UG3 Pilot Clinical Trial
Brief Title: UG3 Pilot Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: HCI177308; UG3CA287109-02 (NIH)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Repeated Text Messages (TM+) (Other): Repeated text messages notifying patients that they may be eligible for Lung Cancer Screening (LCS).
  Interventions: Other: Repeated Text Messages (TM+)
- Repeated Text Messages plus a Conversational Agent (TM+, CA) (Other): Repeated text messages notifying patients that they may be eligible for LCS. In addition to text messages, patients will receive an automated, scripted, and interactive CA.
  Interventions: Other: Repeated Text Messages (TM+); Other: Conversational Agent (CA)
- Repeated Text Messages plus a Video (TM+, Video) (Other): Repeated text messages notifying patients that they may be eligible for LCS. In addition to text messages, patients will receive an educational video sent directly to their cell phone.
  Interventions: Other: Repeated Text Messages (TM+); Other: Educational Video
- Repeated Text Messages plus a Conversational Agent and Video (TM+, CA, Video) (Other): Repeated text messages notifying patients that they may be eligible for LCS. In addition to text messages, patients will receive an educational video sent directly to the patient's cell phone, along with a conversational agent to answer frequently asked LCS questions.
  Additionally, patients will receive an educational video sent directly to the patient's cell phone and a chatbot to answer frequently asked LCS questions.
  Interventions: Other: Repeated Text Messages (TM+); Other: Conversational Agent (CA); Other: Educational Video
- CA/PPN (Other): A conversational agent to answer frequently asked LCS questions. In addition to proactive patient navigation.
  Interventions: Other: Conversational Agent (CA); Other: Proactive Patient Navigation (PPN)
- CA/RPN (Other): A conversational agent to answer frequently asked LCS questions. In addition to reactive patient navigation.
  Interventions: Other: Conversational Agent (CA); Other: Reactive Patient Navigation (RPN)

INTERVENTIONS:
Other: Repeated Text Messages (TM+) — The text message notifies patients that they may be eligible for LCS and provides the patient with a connection to an registered nurse (RN) for LCS eligibility assessment and Shared Decision-Making (SDM) discussion. Response options include YES (to request that the HUB RN call the patient) or STOP (to opt out of any further messages).
  Arms: Repeated Text Messages (TM+); Repeated Text Messages plus a Conversational Agent (TM+, CA); Repeated Text Messages plus a Conversational Agent and Video (TM+, CA, Video); Repeated Text Messages plus a Video (TM+, Video)
Other: Conversational Agent (CA) — The CA is designed to address specific hesitancy factors and barriers to Lung Cancer Screening (LCS). The CA uses a rule-based approach. CAs use a predefined conversation script with a fixed set of possible questions and responses to educate patients regarding the importance of LCS and engage them to be connected with RN for eligibility assessment and SDM.
  Arms: CA/PPN; CA/RPN; Repeated Text Messages plus a Conversational Agent (TM+, CA); Repeated Text Messages plus a Conversational Agent and Video (TM+, CA, Video)
Other: Educational Video — The educational video provides patients with information and answers commonly asked questions about LCS.
  Arms: Repeated Text Messages plus a Conversational Agent and Video (TM+, CA, Video); Repeated Text Messages plus a Video (TM+, Video)
Other: Proactive Patient Navigation (PPN) — Proactive patient navigation enables trained navigators to actively identify and reach out to patients who may need assistance completing LCS, rather than waiting for patients to seek help on their own.
  Arms: CA/PPN
Other: Reactive Patient Navigation (RPN) — Reactive patient navigation makes trained navigators available to those who seek assistance in completing LCS.
  Arms: CA/RPN

SUMMARY:
LungSMART Utah utilizes a Population Health Management (PHM) approach that addresses key barriers to Lung Cancer Screening (LCS) implementation by deploying a centralized Hub infrastructure for eligibility assessment, individualized risk assessment and Shared Decision Making (SDM), LCS referral, and screening completion assistance, thereby increasing LCS reach at scale among Community Health Centers (CHCs) patients across the state of Utah.

DETAILED DESCRIPTION:
LungSMART Utah is a Sequential Multiple Assignment Randomized Trial (SMART) that promotes the reach of lung cancer screening (LCS) among patients who receive medical services at Utah Community Health Centers (CHCs). The study design consists of two sequential stages: an Eligibility Assessment phase to identify and engage individuals at risk to participate in a shared decision-making (SDM) session to assess LCS eligibility, recommendation, and preference, followed by an LCS Completion phase to promote follow-through with recommended screening.

In this pilot trial, 50 current or former tobacco users aged 50-80 who receive medical services at the Mountainlands CHC and have no recorded history of lung cancer and have not participated in a SDM about LCS will be identified for the study. In the Eligibility Assessment Phase, patients will be assessed for LCS eligibility through digital health interventions and, if eligible, will engage with a qualified registered nurse (RN) at a centralized "Hub" for a SDM session, with and be offered a referral for LCS if screening is recommended and preferred. Phase 1 interventions include repeated text messaging (TM+), conversational agent (CA), and educational video (VID) to engage patients in a SDM session. The LCS Completion phase evaluates telehealth interventions designed to address logistical barriers and hesitancy among referred patients in completing LCS. Interventions include CA and either proactive- or reactive-patient navigation (PN) to increase LCS completion among CHC patients. Clinic staff will also be queried to examine if further refinement of research workflow and procedures is needed. Mountainlands CHC has agreed to partner with us to recruit patient participants for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Is currently a patient at Mountainlands CHCs
* Speak English or Spanish
* Current or former male or female smokers
* Age 50-80
* Have a phone that can receive text messages
* Electronic health records indicate they have not opted out of receiving text contact from the clinic

Exclusion Criteria:

* Persons with lung cancer or previous SDM

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Engagement - Lung Cancer Screening (LCS) | up to 3 months from study enrollment
  Survey questions will measure engagement, trustworthiness, acceptability, and usefulness related to all interventions and content.
  LCS text message engagement is measured as a single-item Yes/No question. This outcome measure will report the proportion of subjects who answered Yes to LCS engagement.
Engagement - Shared Decision Making (SDM) | up to 3 months from study enrollment
  Survey questions will measure engagement, trustworthiness, acceptability, and usefulness related to all interventions and content.
  SDM text message engagement is measured as a single-item Yes/No question. This outcome measure will report the proportion of subjects who answered Yes to SDM engagement.

SECONDARY OUTCOMES:
Trustworthiness | up to 3 months from study enrollment
  Survey questions will measure engagement, trustworthiness, acceptability, and usefulness related to all interventions and content.
  Text message trustworthiness is measured by two items that directly ask what made participants trust or not trust the initial text message. This outcome measure will report the proportion of subjects who reported text message trustworthiness.
Acceptability | up to 3 months from study enrollment
  Survey questions will measure engagement, trustworthiness, acceptability, and usefulness related to all interventions and content.
  Acceptability is measured as a composite of 4 dimensions:
  * Frequency: 3 items about text message frequency and call attempt frequency
  * Pace: 2 items about information delivery pace
  * Process: 1 item about technical issues, 2 items regarding improvement suggestions, and 3 open-ended questions about the overall experience
  * Content: 4 Yes/No items about the educational video in the branching logic section.
  This outcome measure will report the proportion of subjects who reported text message acceptability.
Usefulness | up to 3 months from study enrollment
  Survey questions will measure engagement, trustworthiness, acceptability, and usefulness related to all interventions and content.
  Usefulness is measured as a composite of 4 dimensions:
  * Perceived helpfulness: 1 question about the helpfulness of reminder texts, and 1 branching logic question about the helpfulness of additional information provided by the educational video that arrives via text.
  * Confidence outcomes: 1 question measuring confidence in the next steps after shared decision-making
  * Functional utility: 2 questions about opportunities to ask questions/express concerns and suggestions for additional valuable resources
  * Overall utility: 2 closing questions about what worked well and the experience with the program.
  This outcome measure will report the proportion of subjects who reported text message usefulness.

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, Ph.D., Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/ University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Fernandez ME, Schlechter CR, Del Fiol G, Gibson B, Kawamoto K, Siaperas T, Pruhs A, Greene T, Nahum-Shani I, Schulthies S, Nelson M, Bohner C, Kramer H, Borbolla D, Austin S, Weir C, Walker TW, Lam CY, Wetter DW. QuitSMART Utah: an implementation study protocol for a cluster-randomized, multi-level Sequential Multiple Assignment Randomized Trial to increase Reach and Impact of tobacco cessation treatment in Community Health Centers. Implement Sci. 2020 Jan 30;15(1):9. doi: 10.1186/s13012-020-0967-2. PMID 32000812
- [Background] Gibson B, Kramer H, Weir C, Fiol G, Borbolla D, Schlechter CR, Lam C, Nelson M, Bohner C, Schulthies S, Sieperas T, Pruhs A, Nahum-Shani I, Fernandez ME, Wetter DW. Workflow analysis for design of an electronic health record-based tobacco cessation intervention in community health centers. JAMIA Open. 2021 Feb 11;4(3):ooaa070. doi: 10.1093/jamiaopen/ooaa070. eCollection 2021 Jul. PMID 34514352
- [Background] Schlechter CR, Del Fiol G, Lam CY, Fernandez ME, Greene T, Yack M, Schulthies S, Nelson M, Bohner C, Pruhs A, Siaperas T, Kawamoto K, Gibson B, Nahum-Shani I, Walker TJ, Wetter DW. Application of community - engaged dissemination and implementation science to improve health equity. Prev Med Rep. 2021 Oct 26;24:101620. doi: 10.1016/j.pmedr.2021.101620. eCollection 2021 Dec. PMID 34976676
- [Background] Schlechter CR, Del Fiol G, Wetter DW, editors. Rapid and responsive interventions to address covid-19 and promote health equity. Proceedings of the 15th Annual Conference on the Science of Dissemination and Implementation in Health; 2022; Washington, DC, USA.
- [Background] Fritz JM, Del Fiol G, Gibson B, Wetter DW, Solis V, Bennett E, Thackeray A, Goode A, Lundberg K, Romero A, Ford I, Stevens L, Siaperas T, Morales J, Yack M, Greene T. BeatPain Utah: study protocol for a pragmatic randomised trial examining telehealth strategies to provide non-pharmacologic pain care for persons with chronic low back pain receiving care in federally qualified health centers. BMJ Open. 2022 Nov 9;12(11):e067732. doi: 10.1136/bmjopen-2022-067732. PMID 36351735
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] American Cancer Society. Estimated number of deaths by state for 21 cancer sites, 2023. Atlanta, GA: American Cancer Society, 2023.
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Background] US Preventive Services Task Force. Final recommendation statement: lung cancer screening (2013) 2013 [04/04/2021]. Available from: https://www.uspreventiveservicestaskforce.org/uspstf/recommendation/lung-cancer-screeningdecember-2013
- [Background] Zhao H, Xu Y, Huo J, Burks AC, Ost DE, Shih YT. Updated Analysis of Complication Rates Associated With Invasive Diagnostic Procedures After Lung Cancer Screening. JAMA Netw Open. 2020 Dec 1;3(12):e2029874. doi: 10.1001/jamanetworkopen.2020.29874. PMID 33326023
- [Background] Tammemagi MC, Katki HA, Hocking WG, Church TR, Caporaso N, Kvale PA, Chaturvedi AK, Silvestri GA, Riley TL, Commins J, Berg CD. Selection criteria for lung-cancer screening. N Engl J Med. 2013 Feb 21;368(8):728-36. doi: 10.1056/NEJMoa1211776. PMID 23425165
- [Background] Kovalchik SA, Tammemagi M, Berg CD, Caporaso NE, Riley TL, Korch M, Silvestri GA, Chaturvedi AK, Katki HA. Targeting of low-dose CT screening according to the risk of lung-cancer death. N Engl J Med. 2013 Jul 18;369(3):245-254. doi: 10.1056/NEJMoa1301851. PMID 23863051
- [Background] Bach PB, Kattan MW, Thornquist MD, Kris MG, Tate RC, Barnett MJ, Hsieh LJ, Begg CB. Variations in lung cancer risk among smokers. J Natl Cancer Inst. 2003 Mar 19;95(6):470-8. doi: 10.1093/jnci/95.6.470. PMID 12644540
- [Background] Katki HA, Kovalchik SA, Berg CD, Cheung LC, Chaturvedi AK. Development and Validation of Risk Models to Select Ever-Smokers for CT Lung Cancer Screening. JAMA. 2016 Jun 7;315(21):2300-11. doi: 10.1001/jama.2016.6255. PMID 27179989
- [Background] Centers for Medicare and Medicaid Services. Decision memo for screening for lung cancer with low dose computed tomography 2015. Available from: https://www.cms.gov/medicare-coveragedatabase/details/nca-decision-memo.aspx?NCAId=274
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter: what does it mean? (or it takes at least two to tango). Soc Sci Med. 1997 Mar;44(5):681-92. doi: 10.1016/s0277-9536(96)00221-3. PMID 9032835
- [Background] Fedewa SA, Bandi P, Smith RA, Silvestri GA, Jemal A. Lung Cancer Screening Rates During the COVID-19 Pandemic. Chest. 2022 Feb;161(2):586-589. doi: 10.1016/j.chest.2021.07.030. Epub 2021 Jul 21. No abstract available. PMID 34298006
- [Background] Kukhareva PV, Caverly TJ, Li H, Katki HA, Cheung LC, Reese TJ, Del Fiol G, Hess R, Wetter DW, Zhang Y, Taft TY, Flynn MC, Kawamoto K. Inaccuracies in electronic health records smoking data and a potential approach to address resulting underestimation in determining lung cancer screening eligibility. J Am Med Inform Assoc. 2022 Apr 13;29(5):779-788. doi: 10.1093/jamia/ocac020. PMID 35167675
- [Background] Brenner AT, Malo TL, Margolis M, Elston Lafata J, James S, Vu MB, Reuland DS. Evaluating Shared Decision Making for Lung Cancer Screening. JAMA Intern Med. 2018 Oct 1;178(10):1311-1316. doi: 10.1001/jamainternmed.2018.3054. PMID 30105393
- [Background] Tai-Seale M, McGuire TG, Zhang W. Time allocation in primary care office visits. Health Serv Res. 2007 Oct;42(5):1871-94. doi: 10.1111/j.1475-6773.2006.00689.x. PMID 17850524
- [Background] Melzer AC, Golden SE, Ono SS, Datta S, Triplette M, Slatore CG. "We Just Never Have Enough Time". Clinician Views of Lung Cancer Screening Processes and Implementation. Ann Am Thorac Soc. 2020 Oct;17(10):1264-1272. doi: 10.1513/AnnalsATS.202003-262OC. PMID 32497437
- [Background] Wang GX, Baggett TP, Pandharipande PV, Park ER, Percac-Lima S, Shepard JO, Fintelmann FJ, Flores EJ. Barriers to Lung Cancer Screening Engagement from the Patient and Provider Perspective. Radiology. 2019 Feb;290(2):278-287. doi: 10.1148/radiol.2018180212. Epub 2019 Jan 8. PMID 30620258
- [Background] Triplette M, Kross EK, Mann BA, Elmore JG, Slatore CG, Shahrir S, Romine PE, Frederick PD, Crothers K. An Assessment of Primary Care and Pulmonary Provider Perspectives on Lung Cancer Screening. Ann Am Thorac Soc. 2018 Jan;15(1):69-75. doi: 10.1513/AnnalsATS.201705-392OC. PMID 28933940
- [Background] Office of the National Coordinator for Health Information Technology. USCDI Proposed Addition: Smoking Pack-Years 2021 [04/04/2021]. Available from: https://www.healthit.gov/isa/uscdidata/pack-years.
- [Background] Fedewa SA, Kazerooni EA, Studts JL, Smith RA, Bandi P, Sauer AG, Cotter M, Sineshaw HM, Jemal A, Silvestri GA. State Variation in Low-Dose Computed Tomography Scanning for Lung Cancer Screening in the United States. J Natl Cancer Inst. 2021 Aug 2;113(8):1044-1052. doi: 10.1093/jnci/djaa170. PMID 33176362
- [Background] Caverly TJ, Cao P, Hayward RA, Meza R. Identifying Patients for Whom Lung Cancer Screening Is Preference-Sensitive: A Microsimulation Study. Ann Intern Med. 2018 Jul 3;169(1):1-9. doi: 10.7326/M17-2561. Epub 2018 May 29. PMID 29809244
- [Background] Mazzone PJ, Silvestri GA, Souter LH, Caverly TJ, Kanne JP, Katki HA, Wiener RS, Detterbeck FC. Screening for Lung Cancer: CHEST Guideline and Expert Panel Report. Chest. 2021 Nov;160(5):e427-e494. doi: 10.1016/j.chest.2021.06.063. Epub 2021 Jul 13. PMID 34270968
- [Background] Kukhareva P, Martin DK, Warner I, Rodriguez S, Li H, Zhang Y, Caverly T, Del Fiol G, Kawamoto K, editors. Lung cancer screening implementation in primary care using an electronic health recordintegrated shared decision making tool and clinician-facing prompts. AMIA Annu Symp Proc; 2022
- [Background] Cornelius ME, Wang TW, Jamal A, Loretan CG, Neff LJ. Tobacco Product Use Among Adults - United States, 2019. MMWR Morb Mortal Wkly Rep. 2020 Nov 20;69(46):1736-1742. doi: 10.15585/mmwr.mm6946a4. PMID 33211681
- [Background] National Center for Health Statistics. Table A-12a. Age-adjusted percentages (with standard errors) of current cigarette smoking status among adults aged 18 and over, by selected characteristics: United States, 2018. Summary health statistics tables: National Health Interview Survey, 2018 2018. Available from: https://ftp.cdc.gov/pub/Health_Statistics/NCHS/NHIS/SHS/2018_SHS_Table_A-12.pdf
- [Background] Office of Disease Prevention and Health Promotion. Adults who are current smokers: Health People 2020. Available from: https://www.healthypeople.gov/2020/leading-health-indicators/2020-lhitopics/Tobacco/data
- [Background] Doogan NJ, Roberts ME, Wewers ME, Stanton CA, Keith DR, Gaalema DE, Kurti AN, Redner R, Cepeda-Benito A, Bunn JY, Lopez AA, Higgins ST. A growing geographic disparity: Rural and urban cigarette smoking trends in the United States. Prev Med. 2017 Nov;104:79-85. doi: 10.1016/j.ypmed.2017.03.011. Epub 2017 Mar 16. PMID 28315761
- [Background] Roberts ME, Doogan NJ, Kurti AN, Redner R, Gaalema DE, Stanton CA, White TJ, Higgins ST. Rural tobacco use across the United States: How rural and urban areas differ, broken down by census regions and divisions. Health Place. 2016 May;39:153-9. doi: 10.1016/j.healthplace.2016.04.001. Epub 2016 Apr 22. PMID 27107746
- [Background] Roberts ME, Doogan NJ, Stanton CA, Quisenberry AJ, Villanti AC, Gaalema DE, Keith DR, Kurti AN, Lopez AA, Redner R, Cepeda-Benito A, Higgins ST. Rural Versus Urban Use of Traditional and Emerging Tobacco Products in the United States, 2013-2014. Am J Public Health. 2017 Oct;107(10):1554-1559. doi: 10.2105/AJPH.2017.303967. Epub 2017 Aug 17. PMID 28817323
- [Background] Vander Weg MW, Cunningham CL, Howren MB, Cai X. Tobacco use and exposure in rural areas: Findings from the Behavioral Risk Factor Surveillance System. Addict Behav. 2011 Mar;36(3):231-6. doi: 10.1016/j.addbeh.2010.11.005. Epub 2010 Nov 10. PMID 21146318
- [Background] Glei DA, Lee C, Weinstein M. Socioeconomic disparities in U.S. mortality: The role of smoking and alcohol/drug abuse. SSM Popul Health. 2020 Nov 25;12:100699. doi: 10.1016/j.ssmph.2020.100699. eCollection 2020 Dec. PMID 33335972
- [Background] Adler-Milstein J, Holmgren AJ, Kralovec P, Worzala C, Searcy T, Patel V. Electronic health record adoption in US hospitals: the emergence of a digital "advanced use" divide. J Am Med Inform Assoc. 2017 Nov 1;24(6):1142-1148. doi: 10.1093/jamia/ocx080. PMID 29016973
- [Background] Kruse CS, Kristof C, Jones B, Mitchell E, Martinez A. Barriers to Electronic Health Record Adoption: a Systematic Literature Review. J Med Syst. 2016 Dec;40(12):252. doi: 10.1007/s10916-016-0628-9. Epub 2016 Oct 6. PMID 27714560
- [Background] Heisey-Grove DM. Variation In Rural Health Information Technology Adoption And Use. Health Aff (Millwood). 2016 Feb;35(2):365-70. doi: 10.1377/hlthaff.2015.0861. Epub 2016 Jan 20. PMID 26791835
- [Background] Henry J, Pylypchuk Y, Patel V. Electronic Capabilities for Patient Engagement among U.S. Non-Federal Acute Care Hospitals: 2012-2015. 2016 Sep. In: ASTP Health IT Data Brief [Internet]. Washington (DC): Office of the Assistant Secretary for Technology Policy; 2012. 38. Available from http://www.ncbi.nlm.nih.gov/books/NBK612951/ PMID 40127343
- [Background] Senft N, Butler E, Everson J. Growing Disparities in Patient-Provider Messaging: Trend Analysis Before and After Supportive Policy. J Med Internet Res. 2019 Oct 7;21(10):e14976. doi: 10.2196/14976. PMID 31593539
- [Background] Spooner KK, Salemi JL, Salihu HM, Zoorob RJ. eHealth patient-provider communication in the United States: interest, inequalities, and predictors. J Am Med Inform Assoc. 2017 Apr 1;24(e1):e18-e27. doi: 10.1093/jamia/ocw087. PMID 27497797
- [Background] PEW Research Center. Mobile Fact Sheet 2021. Available from: https://www.pewresearch.org/internet/fact-sheet/mobile/.
- [Background] Ten Haaf K, van der Aalst CM, de Koning HJ, Kaaks R, Tammemagi MC. Personalising lung cancer screening: An overview of risk-stratification opportunities and challenges. Int J Cancer. 2021 Jul 15;149(2):250-263. doi: 10.1002/ijc.33578. Epub 2021 May 3. PMID 33783822
- [Background] Nunez ER, Caverly TJ, Zhang S, Glickman ME, Qian SX, Boudreau JH, Slatore CG, Miller DR, Wiener RS. Adherence to Follow-up Testing Recommendations in US Veterans Screened for Lung Cancer, 2015-2019. JAMA Netw Open. 2021 Jul 1;4(7):e2116233. doi: 10.1001/jamanetworkopen.2021.16233. PMID 34236409
- [Background] Tanner NT, Brasher PB, Wojciechowski B, Ward R, Slatore C, Gebregziabher M, Silvestri GA. Screening Adherence in the Veterans Administration Lung Cancer Screening Demonstration Project. Chest. 2020 Oct;158(4):1742-1752. doi: 10.1016/j.chest.2020.04.063. Epub 2020 May 19. PMID 32439505
- [Background] Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. Epidemiol Rev. 2010;32(1):56-69. doi: 10.1093/epirev/mxq004. Epub 2010 Mar 30. PMID 20354039
- [Background] Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD007458. doi: 10.1002/14651858.CD007458.pub3. PMID 24310741
- [Background] Head KJ, Noar SM, Iannarino NT, Grant Harrington N. Efficacy of text messaging-based interventions for health promotion: a meta-analysis. Soc Sci Med. 2013 Nov;97:41-8. doi: 10.1016/j.socscimed.2013.08.003. Epub 2013 Aug 13. PMID 24161087
- [Background] Schwebel FJ, Larimer ME. Using text message reminders in health care services: A narrative literature review. Internet Interv. 2018 Jun 21;13:82-104. doi: 10.1016/j.invent.2018.06.002. eCollection 2018 Sep. PMID 30206523
- [Background] U.S. Department of Health and Human Services. Using Health Text Messages to Improve Consumer Health Knowledge, Behaviors, and Outcomes: An Environmental Scan. Rockville, Maryland: Health Resources and Services Administration. U.S. Department of Health and Human Services: 2014
- [Background] Vodopivec-Jamsek V, de Jongh T, Gurol-Urganci I, Atun R, Car J. Mobile phone messaging for preventive health care. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007457. doi: 10.1002/14651858.CD007457.pub2. PMID 23235643
- [Background] Community Preventive Services Task Force. CPSTF recommends patient navigation services to increase cancer screening and advance health equity. Available from: https://www.thecommunityguide.org/news/cpstf-recommends-patient-navigation-services-increasecancer-screening-advance-health-equity.html
- [Background] Community Preventive Services Task Force. Cancer screening: Interventions engaging community health workers - colorectal cancer. Available from: https://www.thecommunityguide.org/findings/cancer-screening-interventions-engaging-communityhealth-workers-colorectal-cancer.html
- [Background] Community Preventive Services Task Force. Cancer screening: Interventions engaging community health workers - cervical cancer. Available from: https://www.thecommunityguide.org/findings/cancer-screening-interventions-engaging-communityhealth-workers-cervical-cancer.html.
- [Background] Community Preventive Services Task Force. Cancer screening: Interventions engaging community health workers breast cancer. Available from: https://www.thecommunityguide.org/findings/cancerscreening-interventions-engaging-community-health-workers-breast-cancer.html
- [Background] Clarke AR, Goddu AP, Nocon RS, Stock NW, Chyr LC, Akuoko JA, Chin MH. Thirty years of disparities intervention research: what are we doing to close racial and ethnic gaps in health care? Med Care. 2013 Nov;51(11):1020-6. doi: 10.1097/MLR.0b013e3182a97ba3. PMID 24128746
- [Background] Purnell TS, Calhoun EA, Golden SH, Halladay JR, Krok-Schoen JL, Appelhans BM, Cooper LA. Achieving Health Equity: Closing The Gaps In Health Care Disparities, Interventions, And Research. Health Aff (Millwood). 2016 Aug 1;35(8):1410-5. doi: 10.1377/hlthaff.2016.0158. PMID 27503965
- [Background] Health Resources & Services Administration. Health Center Program Uniform Data System (UDS) Program Awardee Data 2021 [02/01/2023]. Available from: https://data.hrsa.gov/tools/datareporting/program-data
- [Background] Xu Y, Gu Z, Zhang Y, He M, Gerber BS, Sadasivam RS, Liu F, Wang Z. Global trends in smoking cessation research from 2002 to 2021: A bibliometric and visual analysis. Prev Med Rep. 2022 Sep 19;30:101991. doi: 10.1016/j.pmedr.2022.101991. eCollection 2022 Dec. PMID 36193091
- [Background] McClure JB, Westbrook E, Curry SJ, Wetter DW. Proactive, motivationally enhanced smoking cessation counseling among women with elevated cervical cancer risk. Nicotine Tob Res. 2005 Dec;7(6):881-9. doi: 10.1080/14622200500266080. PMID 16298723
- [Background] Reitzel LR, Vidrine JI, Businelle MS, Kendzor DE, Costello TJ, Li Y, Daza P, Mullen PD, Velasquez MM, Cinciripini PM, Cofta-Woerpel L, Wetter DW. Preventing postpartum smoking relapse among diverse low-income women: a randomized clinical trial. Nicotine Tob Res. 2010 Apr;12(4):326-35. doi: 10.1093/ntr/ntq001. Epub 2010 Feb 12. PMID 20154055
- [Background] Vidrine JI, Reitzel LR, Figueroa PY, Velasquez MM, Mazas CA, Cinciripini PM, Wetter DW. Motivation and Problem Solving (MAPS): Motivationally Based Skills Training for Treating Substance Use. Cogn Behav Pract. 2013 Nov;20(4):501-516. doi: 10.1016/j.cbpra.2011.11.001. Epub 2011 Dec 8. PMID 33239855
- [Background] Vinci C, Lam C, Schlechter CR, Shono Y, Vidrine JI, Wetter DW. Increasing treatment enrollment among smokers who are not motivated to quit: a randomized clinical trial. Transl Behav Med. 2022 Jan 18;12(1):ibab114. doi: 10.1093/tbm/ibab114. PMID 34424337
- [Background] Wetter DW, Mazas C, Daza P, Nguyen L, Fouladi RT, Li Y, Cofta-Woerpel L. Reaching and treating Spanish-speaking smokers through the National Cancer Institute's Cancer Information Service. A randomized controlled trial. Cancer. 2007 Jan 15;109(2 Suppl):406-13. doi: 10.1002/cncr.22360. PMID 17149758
- [Background] Bui TC, Pineiro B, Vidrine DJ, Wetter DW, Frank-Pearce SG, Vidrine JI. Quitline Treatment Enrollment and Cessation Outcomes Among Smokers Linked With Treatment via Ask-Advise-Connect: Comparisons Among Smokers With and Without HIV. Nicotine Tob Res. 2020 Aug 24;22(9):1640-1643. doi: 10.1093/ntr/ntz227. PMID 31811295
- [Background] Pineiro B, Vidrine DJ, Wetter DW, Hoover DS, Frank-Pearce SG, Nguyen N, Zbikowski SM, Vidrine JI. Implementation of Ask-Advise-Connect in a safety net healthcare system: quitline treatment engagement and smoking cessation outcomes. Transl Behav Med. 2020 Feb 3;10(1):163-167. doi: 10.1093/tbm/iby108. PMID 30476236
- [Background] Pineiro B, Wetter DW, Vidrine DJ, Hoover DS, Frank-Pearce SG, Nguyen N, Zbikowski SM, Williams MB, Vidrine JI. Quitline treatment dose predicts cessation outcomes among safety net patients linked with treatment via Ask-Advise-Connect. Prev Med Rep. 2019 Jan 17;13:262-267. doi: 10.1016/j.pmedr.2019.01.009. eCollection 2019 Mar. PMID 30723660
- [Background] Vidrine JI, Shete S, Cao Y, Greisinger A, Harmonson P, Sharp B, Miles L, Zbikowski SM, Wetter DW. Ask-Advise-Connect: a new approach to smoking treatment delivery in health care settings. JAMA Intern Med. 2013 Mar 25;173(6):458-64. doi: 10.1001/jamainternmed.2013.3751. PMID 23440173
- [Background] Vidrine JI, Shete S, Li Y, Cao Y, Alford MH, Galindo-Talton M, Rabius V, Sharp B, Harmonson P, Zbikowski SM, Miles L, Wetter DW. The Ask-Advise-Connect approach for smokers in a safety net healthcare system: a group-randomized trial. Am J Prev Med. 2013 Dec;45(6):737-41. doi: 10.1016/j.amepre.2013.07.011. PMID 24237916
- [Background] Reese TJ, Schlechter CR, Kramer H, Kukhareva P, Weir CR, Del Fiol G, Caverly T, Hess R, Flynn MC, Taft T, Kawamoto K. Implementing lung cancer screening in primary care: needs assessment and implementation strategy design. Transl Behav Med. 2022 Feb 16;12(2):187-197. doi: 10.1093/tbm/ibab115. PMID 34424342
- [Background] Kawamoto K, Kukhareva PV, Weir C, Flynn MC, Nanjo CJ, Martin DK, Warner PB, Shields DE, Rodriguez-Loya S, Bradshaw RL, Cornia RC, Reese TJ, Kramer HS, Taft T, Curran RL, Morgan KL, Borbolla D, Hightower M, Turnbull WJ, Strong MB, Chapman WW, Gregory T, Stipelman CH, Shakib JH, Hess R, Boltax JP, Habboushe JP, Sakaguchi F, Turner KM, Narus SP, Tarumi S, Takeuchi W, Ban H, Wetter DW, Lam C, Caverly TJ, Fagerlin A, Norlin C, Malone DC, Kaphingst KA, Kohlmann WK, Brooke BS, Del Fiol G. Establishing a multidisciplinary initiative for interoperable electronic health record innovations at an academic medical center. JAMIA Open. 2021 Jul 31;4(3):ooab041. doi: 10.1093/jamiaopen/ooab041. eCollection 2021 Jul. PMID 34345802
- [Background] Chavez-Yenter D, Kimball KE, Kohlmann W, Lorenz Chambers R, Bradshaw RL, Espinel WF, Flynn M, Gammon A, Goldberg E, Hagerty KJ, Hess R, Kessler C, Monahan R, Temares D, Tobik K, Mann DM, Kawamoto K, Del Fiol G, Buys SS, Ginsburg O, Kaphingst KA. Patient Interactions With an Automated Conversational Agent Delivering Pretest Genetics Education: Descriptive Study. J Med Internet Res. 2021 Nov 18;23(11):e29447. doi: 10.2196/29447. PMID 34792472
- [Background] Liebermann E, Taber P, Vega AS, Daly BM, Goodman MS, Bradshaw R, Chan PA, Chavez-Yenter D, Hess R, Kessler C, Kohlmann W, Low S, Monahan R, Kawamoto K, Del Fiol G, Buys SS, Sigireddi M, Ginsburg O, Kaphingst KA. Barriers to family history collection among Spanish-speaking primary care patients: a BRIDGE qualitative study. PEC Innov. 2022 Dec;1:100087. doi: 10.1016/j.pecinn.2022.100087. Epub 2022 Sep 27. PMID 36532299
- [Background] Taber P, Ghani P, Schiffman JD, Kohlmann W, Hess R, Chidambaram V, Kawamoto K, Waller RG, Borbolla D, Del Fiol G, Weir C. Physicians' strategies for using family history data: having the data is not the same as using the data. JAMIA Open. 2020 Oct 8;3(3):378-385. doi: 10.1093/jamiaopen/ooaa035. eCollection 2020 Oct. PMID 34632321
- [Background] Neta G, Glasgow RE, Carpenter CR, Grimshaw JM, Rabin BA, Fernandez ME, Brownson RC. A Framework for Enhancing the Value of Research for Dissemination and Implementation. Am J Public Health. 2015 Jan;105(1):49-57. doi: 10.2105/AJPH.2014.302206. PMID 25393182
- [Background] Judson TJ, Odisho AY, Neinstein AB, Chao J, Williams A, Miller C, Moriarty T, Gleason N, Intinarelli G, Gonzales R. Rapid design and implementation of an integrated patient self-triage and self-scheduling tool for COVID-19. J Am Med Inform Assoc. 2020 Jun 1;27(6):860-866. doi: 10.1093/jamia/ocaa051. PMID 32267928
- [Background] Judson TJ, Odisho AY, Young JJ, Bigazzi O, Steuer D, Gonzales R, Neinstein AB. Implementation of a digital chatbot to screen health system employees during the COVID-19 pandemic. J Am Med Inform Assoc. 2020 Jul 1;27(9):1450-1455. doi: 10.1093/jamia/ocaa130. PMID 32531066
- [Background] McKillop M, South BR, Preininger A, Mason M, Jackson GP. Leveraging conversational technology to answer common COVID-19 questions. J Am Med Inform Assoc. 2021 Mar 18;28(4):850-855. doi: 10.1093/jamia/ocaa316. PMID 33517402
- [Background] Dennis AR, Kim A, Raimi R, Ayabakan S. User reactions to COVID-19 screening chatbots from reputable providers. J Am Med Inform Assoc. 2020 Nov 1;27(11):1727-1731. doi: 10.1093/jamia/ocaa167. PMID 32984890
- [Background] Ford D, Harvey JB, McElligott J, King K, Simpson KN, Valenta S, Warr EH, Walsh T, Debenham E, Teasdale C, Meystre S, Obeid JS, Metts C, Lenert LA. Leveraging health system telehealth and informatics infrastructure to create a continuum of services for COVID-19 screening, testing, and treatment. J Am Med Inform Assoc. 2020 Dec 9;27(12):1871-1877. doi: 10.1093/jamia/ocaa157. PMID 32602884
- [Background] Vidrine JI, Rabius V, Alford MH, Li Y, Wetter DW. Enhancing dissemination of smoking cessation quitlines through T2 translational research: a unique partnership to address disparities in the delivery of effective cessation treatment. J Public Health Manag Pract. 2010 Jul-Aug;16(4):304-8. doi: 10.1097/PHH.0b013e3181cbc500. No abstract available. PMID 20520368
- [Background] Davies P, Walker AE, Grimshaw JM. A systematic review of the use of theory in the design of guideline dissemination and implementation strategies and interpretation of the results of rigorous evaluations. Implement Sci. 2010 Feb 9;5:14. doi: 10.1186/1748-5908-5-14. PMID 20181130
- [Background] Grol RP, Bosch MC, Hulscher ME, Eccles MP, Wensing M. Planning and studying improvement in patient care: the use of theoretical perspectives. Milbank Q. 2007;85(1):93-138. doi: 10.1111/j.1468-0009.2007.00478.x. PMID 17319808
- [Background] Lewis CC, Proctor EK, Brownson RC. Measurement issues in dissemination and implementation research. Dissemination and implementation research in health: Translating science to practice. 2017;2:229-44
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Main C, Moxham T, Wyatt JC, Kay J, Anderson R, Stein K. Computerised decision support systems in order communication for diagnostic, screening or monitoring test ordering: systematic reviews of the effects and cost-effectiveness of systems. Health Technol Assess. 2010 Oct;14(48):1-227. doi: 10.3310/hta14480. PMID 21034668
- [Background] Fillmore CL, Bray BE, Kawamoto K. Systematic review of clinical decision support interventions with potential for inpatient cost reduction. BMC Med Inform Decis Mak. 2013 Dec 17;13:135. doi: 10.1186/1472-6947-13-135. PMID 24344752
- [Background] Reese TJ, Schlechter CR, Potter LN, Kawamoto K, Del Fiol G, Lam CY, Wetter DW. Evaluation of Revised US Preventive Services Task Force Lung Cancer Screening Guideline Among Women and Racial/Ethnic Minority Populations. JAMA Netw Open. 2021 Jan 4;4(1):e2033769. doi: 10.1001/jamanetworkopen.2020.33769. PMID 33433600
- [Background] Ali MK, McKeever Bullard K, Imperatore G, Benoit SR, Rolka DB, Albright AL, Gregg EW. Reach and Use of Diabetes Prevention Services in the United States, 2016-2017. JAMA Netw Open. 2019 May 3;2(5):e193160. doi: 10.1001/jamanetworkopen.2019.3160. PMID 31074808
- [Background] Chambers DA, Azrin ST. Research and services partnerships: partnership: a fundamental component of dissemination and implementation research. Psychiatr Serv. 2013 Jun;64(6):509-11. doi: 10.1176/appi.ps.201300032. PMID 23728600
- [Background] US Department of Health and Human Services. Social determinants of health. Available from: https://health.gov/healthypeople/priority-areas/social-determinants-health.
- [Background] Center for Disease Control and Prevention. Social determinants of health. Available from: https://www.cdc.gov/socialdeterminants/about.html.
- [Background] Syed ST, Gerber BS, Sharp LK. Traveling towards disease: transportation barriers to health care access. J Community Health. 2013 Oct;38(5):976-93. doi: 10.1007/s10900-013-9681-1. PMID 23543372
- [Background] Hadley J. Sicker and poorer--the consequences of being uninsured: a review of the research on the relationship between health insurance, medical care use, health, work, and income. Med Care Res Rev. 2003 Jun;60(2 Suppl):3S-75S; discussion 76S-112S. doi: 10.1177/1077558703254101. PMID 12800687
- [Background] Lurie N, Dubowitz T. Health disparities and access to health. JAMA. 2007 Mar 14;297(10):1118-21. doi: 10.1001/jama.297.10.1118. No abstract available. PMID 17356034
- [Background] Goding Sauer A, Siegel RL, Jemal A, Fedewa SA. Current Prevalence of Major Cancer Risk Factors and Screening Test Use in the United States: Disparities by Education and Race/Ethnicity. Cancer Epidemiol Biomarkers Prev. 2019 Apr;28(4):629-642. doi: 10.1158/1055-9965.EPI-18-1169. PMID 30944145
- [Background] Douthit N, Kiv S, Dwolatzky T, Biswas S. Exposing some important barriers to health care access in the rural USA. Public Health. 2015 Jun;129(6):611-20. doi: 10.1016/j.puhe.2015.04.001. Epub 2015 May 27. PMID 26025176
- [Background] Pruitt SL, Shim MJ, Mullen PD, Vernon SW, Amick BC 3rd. Association of area socioeconomic status and breast, cervical, and colorectal cancer screening: a systematic review. Cancer Epidemiol Biomarkers Prev. 2009 Oct;18(10):2579-99. doi: 10.1158/1055-9965.EPI-09-0135. PMID 19815634
- [Background] Carney PA, O'Malley J, Buckley DI, Mori M, Lieberman DA, Fagnan LJ, Wallace J, Liu B, Morris C. Influence of health insurance coverage on breast, cervical, and colorectal cancer screening in rural primary care settings. Cancer. 2012 Dec 15;118(24):6217-25. doi: 10.1002/cncr.27635. Epub 2012 May 30. PMID 22648383
- [Background] Hiscock R, Bauld L, Amos A, Fidler JA, Munafo M. Socioeconomic status and smoking: a review. Ann N Y Acad Sci. 2012 Feb;1248:107-23. doi: 10.1111/j.1749-6632.2011.06202.x. Epub 2011 Nov 17. PMID 22092035
- [Background] Mendoza JA, Miller CA, Martin KJ, Resnicow K, Iachan R, Faseru B, McDaniels-Davidson C, Deng Y, Martinez ME, Demark-Wahnefried W, Leader AE, Lazovich D, Jensen JD, Briant KJ, Fuemmeler BF. Examining the Association of Food Insecurity and Being Up-to-Date for Breast and Colorectal Cancer Screenings. Cancer Epidemiol Biomarkers Prev. 2022 May 4;31(5):1017-1025. doi: 10.1158/1055-9965.EPI-21-1116. PMID 35247884
- [Background] Doescher MP, Jackson JE. Trends in cervical and breast cancer screening practices among women in rural and urban areas of the United States. J Public Health Manag Pract. 2009 May-Jun;15(3):200-9. doi: 10.1097/PHH.0b013e3181a117da. PMID 19363399
- [Background] Cole AM, Jackson JE, Doescher M. Urban-rural disparities in colorectal cancer screening: cross-sectional analysis of 1998-2005 data from the Centers for Disease Control's Behavioral Risk Factor Surveillance Study. Cancer Med. 2012 Dec;1(3):350-6. doi: 10.1002/cam4.40. Epub 2012 Oct 30. PMID 23342284
- [Background] Kurani SS, McCoy RG, Lampman MA, Doubeni CA, Finney Rutten LJ, Inselman JW, Giblon RE, Bunkers KS, Stroebel RJ, Rushlow D, Chawla SS, Shah ND. Association of Neighborhood Measures of Social Determinants of Health With Breast, Cervical, and Colorectal Cancer Screening Rates in the US Midwest. JAMA Netw Open. 2020 Mar 2;3(3):e200618. doi: 10.1001/jamanetworkopen.2020.0618. PMID 32150271
- [Background] Henry J, Barker W, Kachay L. Electronic Capabilities for Patient Engagement among U.S. Non-Federal Acute Care Hospitals: 2013-2017. 2019 Apr. In: ASTP Health IT Data Brief [Internet]. Washington (DC): Office of the Assistant Secretary for Technology Policy; 2012. 45. Available from http://www.ncbi.nlm.nih.gov/books/NBK610219/ PMID 39680701
- [Background] Goetz Goldberg D, Kuzel AJ, Feng LB, DeShazo JP, Love LE. EHRs in primary care practices: benefits, challenges, and successful strategies. Am J Manag Care. 2012 Feb 1;18(2):e48-54. PMID 22435884
- [Background] Green LA, Potworowski G, Day A, May-Gentile R, Vibbert D, Maki B, Kiesel L. Sustaining "meaningful use" of health information technology in low-resource practices. Ann Fam Med. 2015 Jan-Feb;13(1):17-22. doi: 10.1370/afm.1740. PMID 25583887
- [Background] PEW Research Center. Internet/Broadband Fact Sheet 2021. Available from: https://www.pewresearch.org/internet/fact-sheet/internet-broadband/
- [Background] Kocaballi AB, Berkovsky S, Quiroz JC, Laranjo L, Tong HL, Rezazadegan D, Briatore A, Coiera E. The Personalization of Conversational Agents in Health Care: Systematic Review. J Med Internet Res. 2019 Nov 7;21(11):e15360. doi: 10.2196/15360. PMID 31697237
- [Background] Inkster B, Sarda S, Subramanian V. An Empathy-Driven, Conversational Artificial Intelligence Agent (Wysa) for Digital Mental Well-Being: Real-World Data Evaluation Mixed-Methods Study. JMIR Mhealth Uhealth. 2018 Nov 23;6(11):e12106. doi: 10.2196/12106. PMID 30470676
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Fulmer R, Joerin A, Gentile B, Lakerink L, Rauws M. Using Psychological Artificial Intelligence (Tess) to Relieve Symptoms of Depression and Anxiety: Randomized Controlled Trial. JMIR Ment Health. 2018 Dec 13;5(4):e64. doi: 10.2196/mental.9782. PMID 30545815
- [Background] Harper R, Nicholl P, McTear M, Wallace J, Black L, Kearney P, editors. Automated Phone Capture of Diabetes Patients Readings with Consultant Monitoring via the Web. 15th Annual IEEE International Conference and Workshop on the Engineering of Computer Based Systems (ecbs 2008); 2008 31 March-4 April 2008
- [Background] Levin E, Levin A. Evaluation of spoken dialogue technology for real-time health data collection. J Med Internet Res. 2006 Dec 11;8(4):e30. doi: 10.2196/jmir.8.4.e30. PMID 17213048
- [Background] Rhee H, Allen J, Mammen J, Swift M. Mobile phone-based asthma self-management aid for adolescents (mASMAA): a feasibility study. Patient Prefer Adherence. 2014 Jan 7;8:63-72. doi: 10.2147/PPA.S53504. eCollection 2014. PMID 24470755
- [Background] Joseph DA, DeGroff A. The CDC Colorectal Cancer Control Program, 2009-2015. Prev Chronic Dis. 2019 Dec 5;16:E159. doi: 10.5888/pcd16.190336. No abstract available. PMID 31808418
- [Background] Joseph DA, DeGroff AS, Hayes NS, Wong FL, Plescia M. The Colorectal Cancer Control Program: partnering to increase population level screening. Gastrointest Endosc. 2011 Mar;73(3):429-34. doi: 10.1016/j.gie.2010.12.027. No abstract available. PMID 21353839
- [Background] Hannon PA, Maxwell AE, Escoffery C, Vu T, Kohn M, Leeman J, Carvalho ML, Pfeiffer DJ, Dwyer A, Fernandez ME, Vernon SW, Liang L, DeGroff A. Colorectal Cancer Control Program grantees' use of evidence-based interventions. Am J Prev Med. 2013 Nov;45(5):644-8. doi: 10.1016/j.amepre.2013.06.010. PMID 24139779
- [Background] University of Michigan Center for Health Communications Research. Lung Cancer Screening Risk Calculator (Decision Precision) 2021 [04/03/2021]. Available from: https://screenlc.com/
- [Background] US Preventive Services Task Force. Final recommendation statement: lung cancer screening 2016 [09/23/2018]. Available from: https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementFinal/lun g-cancer-screening.
- [Background] Caverly T. Selecting the best candidates for lung cancer screening. JAMA Intern Med. 2015 Jun;175(6):898-900. doi: 10.1001/jamainternmed.2015.1235. No abstract available. PMID 25844984
- [Background] National Cancer Institute. Lung Cancer Risk Models for Screening 2021 [04/03/2021]. Available from: https://dceg.cancer.gov/tools/risk-assessment/lcrisks
- [Background] Cheung LC, Berg CD, Castle PE, Katki HA, Chaturvedi AK. Life-Gained-Based Versus Risk-Based Selection of Smokers for Lung Cancer Screening. Ann Intern Med. 2019 Nov 5;171(9):623-632. doi: 10.7326/M19-1263. Epub 2019 Oct 22. PMID 31634914
- [Background] Lin GA, Fagerlin A. Shared decision making: state of the science. Circ Cardiovasc Qual Outcomes. 2014 Mar;7(2):328-34. doi: 10.1161/CIRCOUTCOMES.113.000322. Epub 2014 Feb 4. No abstract available. PMID 24496297
- [Background] Landy R, Young CD, Skarzynski M, Cheung LC, Berg CD, Rivera MP, Robbins HA, Chaturvedi AK, Katki HA. Using Prediction Models to Reduce Persistent Racial and Ethnic Disparities in the Draft 2020 USPSTF Lung Cancer Screening Guidelines. J Natl Cancer Inst. 2021 Nov 2;113(11):1590-1594. doi: 10.1093/jnci/djaa211. PMID 33399825
- [Background] Caverly TJ, Hayward RA. Dealing with the Lack of Time for Detailed Shared Decision-making in Primary Care: Everyday Shared Decision-making. J Gen Intern Med. 2020 Oct;35(10):3045-3049. doi: 10.1007/s11606-020-06043-2. Epub 2020 Aug 10. PMID 32779137
- [Background] Haddad DN, Sandler KL, Henderson LM, Rivera MP, Aldrich MC. Disparities in Lung Cancer Screening: A Review. Ann Am Thorac Soc. 2020 Apr;17(4):399-405. doi: 10.1513/AnnalsATS.201907-556CME. PMID 32017612
- [Background] Rivera MP, Katki HA, Tanner NT, Triplette M, Sakoda LC, Wiener RS, Cardarelli R, Carter-Harris L, Crothers K, Fathi JT, Ford ME, Smith R, Winn RA, Wisnivesky JP, Henderson LM, Aldrich MC. Addressing Disparities in Lung Cancer Screening Eligibility and Healthcare Access. An Official American Thoracic Society Statement. Am J Respir Crit Care Med. 2020 Oct 1;202(7):e95-e112. doi: 10.1164/rccm.202008-3053ST. PMID 33000953
- [Background] Community Preventive Services Task Force. Diabetes management: Interventions engaging community health workers. Available from: https://www.thecommunityguide.org/findings/diabetes-managementinterventions-engaging-community-health-workers.html
- [Background] Community Preventive Services Task Force. Diabetes prevention: Interventions engaging community health workers. Available from: https://www.thecommunityguide.org/findings/diabetes-preventioninterventions-engaging-community-health-workers.html
- [Background] Community Preventive Services Task Force. Heart disease and stroke prevention: Interventions engaging community health workers. Available from: https://www.thecommunityguide.org/findings/heart-disease-stroke-prevention-interventionsengaging-community-health-workers.html
- [Background] Abrams DB, Monti PM, Niaura RS, Rohsenow DJ, Colby SM. Interventions for Alcoholics Who Smoke. Alcohol Health Res World. 1996;20(2):111-117. PMID 31798159
- [Background] Michie S, Atkins L, West R. The behaviour change wheel. A guide to designing interventions 1st ed Great Britain: Silverback Publishing. 2014:1003-10
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Marlatt GA, Gordon JR. Relapse Prevention:Maintenance strategies in the treatment of addictive behaviors. New York: Guilford Press; 1985
- [Background] Marlatt G. Relapse prevention: Theoretical rationale and overview of the model. In: Marlatt G, Gordon JR, editors. Relapse prevention: Maintenance strategies in the treatment of addictive behaviors New York: Guilford Press; 1985. p. 3-70
- [Background] Sheeran P, Maki A, Montanaro E, Avishai-Yitshak A, Bryan A, Klein WM, Miles E, Rothman AJ. The impact of changing attitudes, norms, and self-efficacy on health-related intentions and behavior: A meta-analysis. Health Psychol. 2016 Nov;35(11):1178-1188. doi: 10.1037/hea0000387. Epub 2016 Jun 9. PMID 27280365
- [Background] Webb TL, Sheeran P. Does changing behavioral intentions engender behavior change? A meta-analysis of the experimental evidence. Psychol Bull. 2006 Mar;132(2):249-68. doi: 10.1037/0033-2909.132.2.249. PMID 16536643
- [Background] Sheeran P, Wright CE, Avishai A, Villegas ME, Rothman AJ, Klein WMP. Does increasing autonomous motivation or perceived competence lead to health behavior change? A meta-analysis. Health Psychol. 2021 Oct;40(10):706-716. doi: 10.1037/hea0001111. PMID 34881939
- [Background] Rimal RN. Closing the knowledge-behavior gap in health promotion: the mediating role of self-efficacy. Health Commun. 2000;12(3):219-37. doi: 10.1207/S15327027HC1203_01. PMID 10938914
- [Background] Carter-Harris L, Slaven JE 2nd, Monahan PO, Draucker CB, Vode E, Rawl SM. Understanding lung cancer screening behaviour using path analysis. J Med Screen. 2020 Jun;27(2):105-112. doi: 10.1177/0969141319876961. Epub 2019 Sep 24. PMID 31550991
- [Background] Miller WR, Zweben A, DiClemente CC, Rychtarik RG. Motivational Enhancement Therapy Manuel: A Clinical Research Guide for Therapists Training Individuals with Alcohol Abuse and Dependence. Rockville, MD: USDHHS, 1995 Contract No.: 94-3723
- [Background] Bandura A. Toward a Psychology of Human Agency. Perspect Psychol Sci. 2006 Jun;1(2):164-80. doi: 10.1111/j.1745-6916.2006.00011.x. PMID 26151469
- [Background] Marlatt G, Donovan D, editors. Relapse prevention: Maintenance strategies in the treatment of addictive behaviors (2nd edition). New York: Guilford Press; 2005
- [Background] USDHHS. Using Health Text Messages To Improve Consumer Health Knowledge, Behaviors, And Outcomes: An Environmental Scan. Rockville, MD: US Department of Health and Human Services, 2014.
- [Background] Wetter DW. How can we help more smokers engage in evidence-based treatment? Annual Conference of the Utah Cancer Action Network; Salt Lake City, UT2017
- [Background] McBrien KA, Ivers N, Barnieh L, Bailey JJ, Lorenzetti DL, Nicholas D, Tonelli M, Hemmelgarn B, Lewanczuk R, Edwards A, Braun T, Manns B. Patient navigators for people with chronic disease: A systematic review. PLoS One. 2018 Feb 20;13(2):e0191980. doi: 10.1371/journal.pone.0191980. eCollection 2018. PMID 29462179
- [Background] Peart A, Lewis V, Brown T, Russell G. Patient navigators facilitating access to primary care: a scoping review. BMJ Open. 2018 Mar 17;8(3):e019252. doi: 10.1136/bmjopen-2017-019252. PMID 29550777
- [Background] Valaitis RK, Carter N, Lam A, Nicholl J, Feather J, Cleghorn L. Implementation and maintenance of patient navigation programs linking primary care with community-based health and social services: a scoping literature review. BMC Health Serv Res. 2017 Feb 6;17(1):116. doi: 10.1186/s12913-017-2046-1. PMID 28166776
- [Background] Correa-Fernandez V, Diaz-Toro EC, Reitzel LR, Guo L, Chen M, Li Y, Calo WA, Shih YT, Wetter DW. Combined treatment for at-risk drinking and smoking cessation among Puerto Ricans: A randomized clinical trial. Addict Behav. 2017 Feb;65:185-192. doi: 10.1016/j.addbeh.2016.10.009. Epub 2016 Oct 22. PMID 27825036
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People to Change Addictive Behavior. New York: The Guildford Press; 1991
- [Background] Miller WR, Rollnick S. Motivational Interviewing (2nd edition). New York: The Guilford Press; 2002
- [Background] Witkiewitz K, Marlatt GA. Relapse prevention for alcohol and drug problems: that was Zen, this is Tao. Am Psychol. 2004 May-Jun;59(4):224-35. doi: 10.1037/0003-066X.59.4.224. PMID 15149263
- [Background] CDC. Telephone Quitlines: A Resource for Development, Implementation, and Evaluation. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Office of Smoking and Health, Final Edition,, 2004 September Report No
- [Background] Moyers TB, Martin T, Manuel JK, Miller WR. The Motivational Interviewing Treatment Integrity (MITI) Code: Version 2.0. nd
- [Background] Muehlen Mz, Recker J. How much language is enough? Theoretical and practical use of the business process modeling notation. In: Bubenko J, Krogstie J, Pastor O, Pernici B, Rolland C, Sølvberg A, editors. Seminal Contributions to Information Systems Engineering: 25 Years of CAiSE. Berlin, Heidelberg: Springer Berlin Heidelberg; 2013. p. 429-43
- [Background] Ramos-Merino M, Alvarez-Sabucedo LM, Santos-Gago JM, Sanz-Valero J. A BPMN Based Notation for the Representation of Workflows in Hospital Protocols. J Med Syst. 2018 Aug 29;42(10):181. doi: 10.1007/s10916-018-1034-2. PMID 30155797
- [Background] Griner D, Smith TB. Culturally adapted mental health intervention: A meta-analytic review. Psychotherapy (Chic). 2006 Winter;43(4):531-48. doi: 10.1037/0033-3204.43.4.531. PMID 22122142
- [Background] Orlandi MA, Freeman H. Smoking control interventions for special populations: Beyond cultural sensitivity. In: Cocores J, editor. The Clinical Management of Nicotine Dependence. New York: Springer-Verlag; 1991. p. 36-46
- [Background] Schinke S, Orlandi MA, Schilling R, Botvin G, Gilchrist L, Landers C. Tobacco use by American Indian and Alaska native people: Risks, psychosocial factors, and preventive intervention. J Alcohol Drug Educ. 1990;35(2):1-12
- [Background] Minkler M, Wallerstein N. Introduction to Community-Based Participatory Research. In: Minkler M, Wallerstein N, editors. Community based participatory research for health. San Francisco, CA: JosseyBass; 2003. p. 3-26
- [Background] Brislin R, Lonner W, Thorndike E. Cross-Cultural Research Methods. New York: Wiley; 1973.
- [Background] Castro Y, Fernandez ME, Strong LL, Stewart DW, Krasny S, Hernandez Robles E, Heredia N, Spears CA, Correa-Fernandez V, Eakin E, Resnicow K, Basen-Engquist K, Wetter DW. Adaptation of a counseling intervention to address multiple cancer risk factors among overweight/obese Latino smokers. Health Educ Behav. 2015 Feb;42(1):65-72. doi: 10.1177/1090198114560019. Epub 2014 Dec 19. PMID 25527143
- [Background] Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: defined and demystified. Ethn Dis. 1999 Winter;9(1):10-21. PMID 10355471
- [Background] Sinicrope PS, Koller KR, Prochaska JJ, Hughes CA, Bock MJ, Decker PA, Flanagan CA, Merritt ZT, Meade CD, Willetto AL, Resnicow K, Thomas TK, Patten CA. Social Media Intervention to Promote Smoking Treatment Utilization and Cessation Among Alaska Native People Who Smoke: Protocol for the Connecting Alaska Native People to Quit Smoking (CAN Quit) Pilot Study. JMIR Res Protoc. 2019 Nov 22;8(11):e15155. doi: 10.2196/15155. PMID 31755867
- [Background] Patten CA, Lando H, Resnicow K, Decker PA, Smith CM, Hanza MM, Burhansstipanov L, Scott M. Developing health communication messaging for a social marketing campaign to reduce tobacco use in pregnancy among Alaska Native women. J Commun Healthc. 2018;11(4):252-262. doi: 10.1080/17538068.2018.1495929. Epub 2018 Jul 16. PMID 31548863
- [Background] Flores G. Culture and the patient-physician relationship: achieving cultural competency in health care. J Pediatr. 2000 Jan;136(1):14-23. doi: 10.1016/s0022-3476(00)90043-x. No abstract available. PMID 10636968
- [Background] Huerta EE, Macario E. Communicating health risk to ethnic groups: reaching Hispanics as a case study. J Natl Cancer Inst Monogr. 1999;(25):23-6. doi: 10.1093/oxfordjournals.jncimonographs.a024202. No abstract available. PMID 10854453
- [Background] (LCV) LCV. Providing Quality Health Care Services to Immigrant Latino Populations in North Carolina: A Working Conference 1999 [cited 2007 January 19]. Available from: http://www.hhcc.arealahec.dst.nc.us/conferenceproceedings.htm
- [Background] Marin G. AIDS prevention among Hispanics: needs, risk behaviors, and cultural values. Public Health Rep. 1989 Sep-Oct;104(5):411-5. PMID 2508169
- [Background] Castro Y, Vinci C, Heppner WL, Cano MA, Correa-Fernandez V, Wetter DW. Revisiting the Relationship Between Acculturation and Smoking Cessation Among Mexican Americans. Ann Behav Med. 2019 Mar 1;53(3):211-222. doi: 10.1093/abm/kay029. PMID 29746621
- [Background] Fennell BS, Pineiro B, Vidrine DJ, Frank-Pearce SG, Wetter DW, Simmons VN, Vidrine JI. Ask-Advise-Connect: Differential Enrollment and Smoking Cessation Outcomes Between Primary Care Patients Who Received Quitline-Delivered Treatment in Spanish vs English. Ann Fam Med. 2022 Nov-Dec;20(6):519-525. doi: 10.1370/afm.2878. PMID 36443074
- [Background] Vinci C, Guo L, Spears CA, Li L, Correa-Fernandez V, Etcheverry PE, Lam CY, Hoover DS, Wetter DW. Socioeconomic indicators as predictors of smoking cessation among Spanish-Speaking Mexican Americans. Ethn Health. 2019 Oct;24(7):841-853. doi: 10.1080/13557858.2017.1373074. Epub 2017 Sep 1. PMID 28859518
- [Background] Castro Y, Businelle MS, Correa-Fernandez V, Kendzor DE, Mazas CA, Cofta-Woerpel L, Wetter DW. Associations between indicators of acculturation and tobacco dependence among Spanish-speaking Latino smokers. Addict Behav. 2012 Oct;37(10):1101-8. doi: 10.1016/j.addbeh.2012.05.003. Epub 2012 May 24. PMID 22688345
- [Background] Castro Y, Reitzel LR, Businelle MS, Kendzor DE, Mazas CA, Li Y, Cofta-Woerpel L, Wetter DW. Acculturation differentially predicts smoking cessation among Latino men and women. Cancer Epidemiol Biomarkers Prev. 2009 Dec;18(12):3468-75. doi: 10.1158/1055-9965.EPI-09-0450. PMID 19959697
- [Background] Hays PA. Seeing the forest and the trees: The complexities of culture in practice2001.
- [Background] Betancourt JR, Green AR, Carrillo JE. Cultural competence in health care: Emerging frameworks and practical approaches: Commonwealth Fund, Quality of Care for Underserved Populations New York, NY; 2002
- [Background] Del Fiol G, Kohlmann W, Bradshaw RL, Weir CR, Flynn M, Hess R, Schiffman JD, Nanjo C, Kawamoto K. Standards-Based Clinical Decision Support Platform to Manage Patients Who Meet Guideline-Based Criteria for Genetic Evaluation of Familial Cancer. JCO Clin Cancer Inform. 2020 Jan;4:1-9. doi: 10.1200/CCI.19.00120. PMID 31951474
- [Background] Kaphingst KA, Kohlmann W, Chambers RL, Goodman MS, Bradshaw R, Chan PA, Chavez-Yenter D, Colonna SV, Espinel WF, Everett JN, Gammon A, Goldberg ER, Gonzalez J, Hagerty KJ, Hess R, Kehoe K, Kessler C, Kimball KE, Loomis S, Martinez TR, Monahan R, Schiffman JD, Temares D, Tobik K, Wetter DW, Mann DM, Kawamoto K, Del Fiol G, Buys SS, Ginsburg O; BRIDGE research team. Comparing models of delivery for cancer genetics services among patients receiving primary care who meet criteria for genetic evaluation in two healthcare systems: BRIDGE randomized controlled trial. BMC Health Serv Res. 2021 Jun 2;21(1):542. doi: 10.1186/s12913-021-06489-y. PMID 34078380
- [Background] Bradshaw RL, Kawamoto K, Kaphingst KA, Kohlmann WK, Hess R, Flynn MC, Nanjo CJ, Warner PB, Shi J, Morgan K, Kimball K, Ranade-Kharkar P, Ginsburg O, Goodman M, Chambers R, Mann D, Narus SP, Gonzalez J, Loomis S, Chan P, Monahan R, Borsato EP, Shields DE, Martin DK, Kessler CM, Del Fiol G. GARDE: a standards-based clinical decision support platform for identifying population health management cohorts. J Am Med Inform Assoc. 2022 Apr 13;29(5):928-936. doi: 10.1093/jamia/ocac028. PMID 35224632
- [Background] Tudor Car L, Dhinagaran DA, Kyaw BM, Kowatsch T, Joty S, Theng YL, Atun R. Conversational Agents in Health Care: Scoping Review and Conceptual Analysis. J Med Internet Res. 2020 Aug 7;22(8):e17158. doi: 10.2196/17158. PMID 32763886
- [Background] United States Census Bureau. National Demographic Analysis Tables: 2020. Available from: https://www.census.gov/data/tables/2020/demo/popest/2020-demographic-analysis-tables.html
- [Background] Dharod A, Bellinger C, Foley K, Case LD, Miller D. The Reach and Feasibility of an Interactive Lung Cancer Screening Decision Aid Delivered by Patient Portal. Appl Clin Inform. 2019 Jan;10(1):19-27. doi: 10.1055/s-0038-1676807. Epub 2019 Jan 9. PMID 30625501
- [Background] Kinsinger LS, Anderson C, Kim J, Larson M, Chan SH, King HA, Rice KL, Slatore CG, Tanner NT, Pittman K, Monte RJ, McNeil RB, Grubber JM, Kelley MJ, Provenzale D, Datta SK, Sperber NS, Barnes LK, Abbott DH, Sims KJ, Whitley RL, Wu RR, Jackson GL. Implementation of Lung Cancer Screening in the Veterans Health Administration. JAMA Intern Med. 2017 Mar 1;177(3):399-406. doi: 10.1001/jamainternmed.2016.9022. PMID 28135352
- [Background] Benkeser D, Diaz I, Luedtke A, Segal J, Scharfstein D, Rosenblum M. Improving precision and power in randomized trials for COVID-19 treatments using covariate adjustment, for binary, ordinal, and time-to-event outcomes. Biometrics. 2021 Dec;77(4):1467-1481. doi: 10.1111/biom.13377. Epub 2020 Oct 11. PMID 32978962
- [Background] Almirall D, Collins LM, Murphy SA. Introduction to adaptive interventions and SMART study design principles. COPTR Workshop on Adaptive Interventions 2011
- [Background] Bierman KL, Nix RL, Maples JJ, Murphy SA; Conduct Problems Prevention Research Group. Examining clinical judgment in an adaptive intervention design: The fast track program. J Consult Clin Psychol. 2006 Jun;74(3):468-81. doi: 10.1037/0022-006X.74.3.468. PMID 16822104
- [Background] McKay JR. Is there a case for extended interventions for alcohol and drug use disorders? Addiction. 2005 Nov;100(11):1594-610. doi: 10.1111/j.1360-0443.2005.01208.x. PMID 16277622
- [Background] Lei H, Nahum-Shani I, Lynch K, Oslin D, Murphy SA. A "SMART" design for building individualized treatment sequences. Annu Rev Clin Psychol. 2012;8:21-48. doi: 10.1146/annurev-clinpsy-032511-143152. Epub 2011 Dec 12. PMID 22224838
- [Background] Dawson R, Lavori PW. Efficient design and inference for multistage randomized trials of individualized treatment policies. Biostatistics. 2012 Jan;13(1):142-52. doi: 10.1093/biostatistics/kxr016. Epub 2011 Jul 16. PMID 21765180
- [Background] Lavori PW, Dawson R, Rush AJ. Flexible treatment strategies in chronic disease: clinical and research implications. Biol Psychiatry. 2000 Sep 15;48(6):605-14. doi: 10.1016/s0006-3223(00)00946-x. PMID 11018231
- [Background] Murphy SA. An experimental design for the development of adaptive treatment strategies. Stat Med. 2005 May 30;24(10):1455-81. doi: 10.1002/sim.2022. PMID 15586395
- [Background] International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonised Tripartite Guideline: Statistical Principles for Clinical Trials E9. London, England: European Medicines Agency, 1998
- [Background] Tibshirani R. Regression shrinkage and selection via the lasso. Journal of the Royal Statistical Society: Series B (Methodological). 1996;58(1):267-88. doi: https://doi.org/10.1111/j.2517- 6161.1996.tb02080.x
- [Background] Tsiatis AA. Dynamic treatment regimes : statistical methods for precision medicine. Boca Raton: CRC Press/Taylor & Francis Group,; 2020.
- [Background] Frangakis CE, Rubin DB. Principal stratification in causal inference. Biometrics. 2002 Mar;58(1):21-9. doi: 10.1111/j.0006-341x.2002.00021.x. PMID 11890317